CLINICAL TRIAL: NCT04519411
Title: Transpulmonary Pressure Measurements in Intubated Children With Covid-19 Respiratory Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to a very low rate of children with COVID-19 pneumonia that required endotracheal intubation, resulting in no eligible subjects to enroll.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen J. Gleich, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-003743
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intubated pediatric patients with COVID-19 respiratory failure (Experimental)
  Interventions: Diagnostic Test: Transpulmonary pressure measurements

INTERVENTIONS:
Diagnostic Test: Transpulmonary pressure measurements — Transpulmonary pressure measurements

SUMMARY:
The purpose of this study is to gather information to help doctors understand how Covid-19 affects the lungs in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-17 years of age, 10 kg or greater, with suspected or confirmed Covid-19 respiratory failure requiring endotracheal intubation and mechanical ventilation admitted to Mayo Clinic Hospital, St. Mary's Campus Pediatric Intensive Care Unit.

Exclusion Criteria:

* Patients <10 kg
* Patients with pre-existing chronic mechanical ventilation (chronic respiratory failure)
* Patients with known esophageal disease (strictures, known esophageal anatomic abnormalities)
* Patients with severe coagulopathy (for which placement of esophageal balloon or other gastric tube via nose or mouth is contraindicated)
* Patients who are pregnant (as determined by standard pregnancy testing criteria for Pediatric ICU admission).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Transpulmonary pressure | Through study complication, usually 2 weeks
  Numerical data

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Gleich, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials